CLINICAL TRIAL: NCT06281483
Title: Efficacy of Platelet-rich Plasma Versus Platelet-rich Fibrin Versus Conventional Treatment in Chronic Non-healing Skin Ulcers: a Comparative Study
Brief Title: PRP Versus PRF Versus Conventional Treatment in Chronic Non-healing Skin Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Collaborators: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed Aboshabana Hussein Mohamed, Assistant Lecturer of Dermatology and Venereology, Kafrelsheikh University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: APCs in chronic skin ulcers
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Chronic Non-healing Skin Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PRP / Group A (Active Comparator): 12 patient
  Interventions: Other: platelet-rich plasma
- PRF / Group B (Active Comparator): 12 patient
  Interventions: Other: platelet-rich fibrin
- Group C (the control group) (Active Comparator): 12 patient
  Interventions: Other: Surgical debridement, normal saline washing and dressing coverage

INTERVENTIONS:
Other: platelet-rich plasma — Under aseptic conditions, 20 mL of whole blood will be withdrawn from each patient and will be collected in the centrifuge tube prefilled with Anticoagulant Citrate Dextrose (1.5 mL each). A two-stage centrifugation process (double-spin method) will be employed for the preparation of PRP. The first spin is at 100 relative centrifugal force (RCF) (g) for 10 min, while the second spin is at 400 RCF for 10 min. PRP will be injected into the base of the ulcer and the surrounding skin. Group A: will receive treatment that will include PRP application, conventional debridement, and dressing coverage. Sessions will be repeated weekly for a maximum of eight sessions.
  Arms: PRP / Group A
Other: platelet-rich fibrin — 20 ml blood will be drawn from each patient by venipuncture under aseptic precautions in four sterile glass tubes of 5-ml capacity without anticoagulant and immediately centrifuged. A single stage centrifugation process, that is (200 g for 8 min), has been found to produce a fibrin clot with the highest platelet and WBC count and highest overall cumulative growth factor yield. Group B: will receive treatment that will include PRF application, conventional debridement, and dressing coverage. Sessions will be repeated weekly for a maximum of eight sessions.
  Arms: PRF / Group B
Other: Surgical debridement, normal saline washing and dressing coverage — Each patient will receive the same conventional debridement and dressing coverage (After opening the bandage, the ulcer will be irrigated with normal saline and will be prepared for debridement as required to remove dead tissues and hyperkeratotic skin. Then, a second wash with normal saline will be done to remove any debris), but without any PRP nor PRF application.
  Arms: Group C (the control group)

SUMMARY:
To compare the therapeutic efficacy of PRP and PRF: two relatively newer modalities in the management of chronic non-healing ulcers versus conventional treatment.

DETAILED DESCRIPTION:
An ulcer is a breach in the continuity of skin, epithelium or mucous membrane caused by sloughing out of inflamed necrotic tissue. Chronic ulcers are formed because of the failure in the orderly process that produces anatomic and functional integrity. Ulcers are considered chronic if they show no tendency to heal after six weeks of appropriate treatment or those that have not fully healed after 12 months.

Despite greater understanding of the biology of wound healing over the past 20 years, some chronic wounds, such as venous leg ulcers, pressure ulcers, and diabetic foot ulcers, are recalcitrant to healing.

In addition to local wound-related factors (eg, ischemia, infection) and patient related factors (eg, diabetes, old age, obesity, malnutrition) that can impair healing, reduction in tissue growth factors, an imbalance between proteolytic enzymes and their inhibitors, and the presence of senescent cells seem to be particularly important in chronic wounds.

Regardless of the underlying etiology, non-healing ulcers tend to have chronic pain, discharge, sleep impairment, and subsequent adverse repercussions in quality of life and productivity, and impose a huge economic burden on the medical system.

In the United States, chronic ulcers including decubitus, vascular, inflammatory, and rheumatologic subtypes affect 6 million people, with increasing numbers anticipated in a growing elderly and diabetic populations.

Venous, arterial, and neuropathic ulcers account for up to 90 percent of ulcers. In a survey study in which wound care professionals in Germany reported the etiologies of chronic leg ulcers in over 31,000 patients, venous insufficiency, arterial insufficiency, and mixed venous and arterial insufficiency accounted for 48, 15, and 18 percent of chronic ulcers, respectively. There are multiple less common causes of ulcers, including physical injury, infection, vasculopathy, pyoderma gangrenosum, panniculitis, malignancy, medications.

The characteristics and difficulties in healing chronic ulcers lie in the lack of an adequate blood supply, long-term repeated inflammatory stimulation in the surrounding tissues, and the presence of a dead cavity. For chronic ulcers, the key is to determine the cause, determine the factors that affect the healing process, and create an environment suitable for healing to effectively treat the wound.

Current therapies include debridement, offloading, etc. However, the response to treatment is often poor, and the outcome is disappointing. These wounds place the limb at the risk of infection and amputation and also puts the patients at risk of mortality.

Chronic ulcers are known to have reduced levels of platelet-derived growth factor, basic fibroblast growth factor, epidermal growth factor, and transforming growth factorβ compared with acute wounds. It has been suggested that growth factors may become trapped by extracellular matrix molecules or may be degraded by proteases to an excessive degree, resulting in non-healing.

Many of the growth factors released from platelets play an important role in the wound-healing process, and topical application of concentrated activated platelets can stimulate wound healing in situations where standard wound care treatments are ineffective.

Platelet-rich concentrates, known as autologous platelet concentrates (APCs), have garnered significant attention in recent years and demonstrate remarkable potential in wound treatment.

Previous studies have shown that activated platelets undergo exocytosis of intracellular granules containing growth factors such as platelet-derived growth factor (PDGF), transforming growth factor-β (TGF-β), epidermal growth factor (EGF), vascular endothelial growth factor (VEGF), and insulin like growth factor (IGF). These growth factors contribute to wound healing by promoting regeneration and wound repair, thereby elucidating the efficacy of APCs therapy in skin regeneration, acne scar treatment, and enhanced wound healing.

APCs can be further classified into platelet-rich plasma (PRP) and platelet-rich fibrin (PRF) based on distinct preparation processes, each with varied clinical applications. PRP, as the first-generation platelet concentrate, is plasma with a high platelet concentration obtained through specific centrifugation of fresh whole blood. PRP contains platelet concentrations four to five times higher than that of whole blood. It has demonstrated positive effects on bone regeneration and wound healing.

PRF, on the other hand, as the second-generation platelet concentrate, exhibits a slow release of growth factors, thereby prolonging their action.

APCs has a greater capacity to modulate the local microenvironment and expedite tissue regeneration. It has also been observed to alleviate pain, accelerate epithelization, and facilitate complete wound healing.

Currently, PRP and PRF, whose therapeutic value is equal to that of stem cells, are currently one of the most promising therapy agents in regenerative medicine. They are increasingly being used in different areas of medicine including aesthetic dermatology, orthopedics, sports medicine and surgery.

Because of the lack of sufficient literature, our study aimed to compare the efficacy of PRP versus PRF versus conventional treatment as a relatively newer modalities in the management of chronic non-healing skin ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with cutaneous ulcers greater than six weeks of duration and a size ranging between 0.5 and 10 cm, having a normal platelet count and hemoglobin >10 gm%.

Exclusion Criteria:

* Patients with known bleeding disorders, and/or on oral anticoagulant therapy, uncontrolled diabetes, proven malignancy.
* Patients who are pregnant or lactating.
* Patients with actively infected ulcers, clinically defined by purulent discharge, green discoloration or fever, or positive culture, ulcers with exposed bone with no underlying granulation tissue, HIV, HCV, HBV patients.
* Patients who are with unrealistic expectations and unwilling to give consent for treatment or photography.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Objective assessment of ulcer size for effectiveness, using Image J software. | Four months of follow up after eight sessions of treatment (six months total)
  Photographs will be obtained at baseline, one month after and at end of eight sessions (two months) with a Nikon D3300 AF-P 18-55 VR 24.2 Megapixels® digital camera and will be standardized for light and distance from the ulcer.
Pain assessment | Four months of follow up after eight sessions of treatment (six months total)
  Pain assessment will be done using Visual analogue scale (scale: 0-10).The Visual analogue scale provides a continuous scale for subjective magnitude estimation and consists of a straight line, the limits of which carry a verbal description of each extreme of the pain to be evaluated. The line is usually 10 cm long and vertical. The Visual analogue scale is often used to evaluate the analgesic properties of various treatments and accomplishes this by measuring either pain relief or pain severity.
Any adverse effects related to treatment modality | Four months of follow up after eight sessions of treatment (six months total)
  Any adverse effects related to therapy will be recorded immediately at each sitting and statistically analyzed for comparison between groups of trial.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Mahmoud Diab, Professor, Study Chair — Ain Shams University
Locations (1):
- Badr Hospital - Helwan University and Kafrelseikh University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badran Z, Abdallah MN, Torres J, Tamimi F. Platelet concentrates for bone regeneration: Current evidence and future challenges. Platelets. 2018 Mar;29(2):105-112. doi: 10.1080/09537104.2017.1327656. Epub 2017 Jun 26. PMID 28649897
- [Background] Chen J, Wan Y, Lin Y, Jiang H. Platelet-rich fibrin and concentrated growth factors as novel platelet concentrates for chronic hard-to-heal skin ulcers: a systematic review and Meta-analysis of randomized controlled trials. J Dermatolog Treat. 2022 Mar;33(2):613-621. doi: 10.1080/09546634.2020.1773386. Epub 2020 Jun 1. PMID 32441168
- [Background] Dashore S, Chouhan K, Nanda S, Sharma A. Platelet-Rich Fibrin, Preparation and Use in Dermatology. Indian Dermatol Online J. 2021 Nov 25;12(Suppl 1):S55-S65. doi: 10.4103/idoj.idoj_282_21. eCollection 2021 Nov. PMID 34976881
- [Background] Evans AG, Ivanic MG, Botros MA, Pope RW, Halle BR, Glassman GE, Genova R, Al Kassis S. Rejuvenating the periorbital area using platelet-rich plasma: a systematic review and meta-analysis. Arch Dermatol Res. 2021 Nov;313(9):711-727. doi: 10.1007/s00403-020-02173-z. Epub 2021 Jan 12. PMID 33433716
- [Background] Muthuprabakaran K, Pai VV, Ahmad S, Shukla P. A cross-sectional analysis of the effects of various centrifugation speeds and inclusion of the buffy coat in platelet-rich plasma preparation. Indian J Dermatol Venereol Leprol. 2021 Nov-Dec;87(6):792-799. doi: 10.25259/IJDVL_1050_20. PMID 34245527